CLINICAL TRIAL: NCT06857968
Title: Improving Opioid Use Disorder Treatment Engagement Using Mobile Mindfulness in Childhood Trauma Survivors
Brief Title: Mobile Mindfulness Training (mMT) for People in Medication Treatment of Opioid Use Disorder (MOUD)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Amy Meadows (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Amy Meadows, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 97193; K23DA054309 (NIH)
Record Dates: First submitted 2025-03-03; First posted 2025-03-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-06

CONDITIONS: Opioid Use Disorder
Keywords: opioid use disorder; mindfulness; childhood trauma; treatment
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual First (Active Comparator): This is a crossover trial. Participants in this study arm will have 30 days of treatment as usual then a 14 day washout and then 30 days of mobile mindfulness training
  Interventions: Behavioral: Mobile Mindfulness Training
- Mobile Mindfulness First (Experimental): This is a crossover trial. Participants in this arm will have 30 days of mobile mindfulness training first then a 14 day washout and then 30 days of treatment as ususal.
  Interventions: Behavioral: Mobile Mindfulness Training

INTERVENTIONS:
Behavioral: Mobile Mindfulness Training — Participants will be instructed to complete a mobile application-based mindfulness training daily for 30 days.
  Other Names: Headspace

SUMMARY:
The goal of this clinical trial is to learn if mobile mindfulness training can help people in treatment for opioid use disorder. The main questions it aims to answer are:

* Will people with opioid use disorder and childhood trauma use mobile mindfulness training?
* Will mobile mindfulness training help people with opioid use disorder and childhood trauma have decreased markers of psychological stress?

Participants will:

Be given access to mobile mindfulness training and encouragement to use it daily for 30 days.

Keep a diary of how often mobile mindfulness training is used. Visit the clinic four times to measure stress levels, including written rating scales, blood work, and heart rate tests.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with Opioid Use Disorder (per DSM5 criteria)
* Currently enrolled in treatment for Opioid Use Disorder at a clinic affiliated with UKHealthCare or University of Kentucky
* On a stable dose of buprenorphine, buprenorphine/naloxone, or naloxone (i.e., at least 30 days post-induction and on a stable dose for 30 days)
* Able to read and understand English
* Have a history of childhood trauma as measured by the Adverse Childhood Experiences scale and/or Childhood Trauma Questionnaire.

Exclusion Criteria:

* Currently taking a beta-blocker, calcium-channel blocker, antiarrhythmic, corticosteroid, or immune modulator medication
* Uncontrolled acute or chronic health conditions (e.g., active infections, autoimmune conditions, cancer undergoing active treatment)
* Current or expected pregnancy
* Current mindfulness practice (i.e., participant reports practicing mindfulness for 10 minutes or more per week)
* Primary psychotic illness
* Diagnosis of a disorder known to interfere with neurocognitive function (e.g., estimated full scale IQ below 70 or diagnosis of dementia)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Access | 75 days after enrollment
  Proportion of enrolled participants who access the online mobile mindfulness training (mMT) application at least once.
Proportion of Acceptability | 75 days after enrollment
  Proportion of enrolled active condition participants who report using the online mobile mindfulness training application at least 25 times in 30 days.

SECONDARY OUTCOMES:
Change in Trauma Symptoms | 180 days after enrollment
  Self-reported changes in trauma symptoms as measured by the Post-Traumatic Stress Disorder Checklist for Diagnostic and Statistical Manual-5 between baseline and 180 days after enrollment. Items are summed to provide a total severity score (range 0-80) with higher scores indicating more symptoms of trauma.
Change in Mindfulness | 180 days after enrollment
  Self-reported changes in mindfulness between as measured by the Five Factor Mindfulness Questionnaire. The Five Factor Mindfulness Questionnaire (FFMQ). It examines 5 key domains of mindfulness: observing, describing, acting with awareness, nonjudging of inner experience, and nonreactivity to inner experience. Scores range from 39 to 195, with higher scores indicating greater tendency to be mindful.

OTHER OUTCOMES:
Change in Heart Rate Variability | 180 days after enrollment
  Change in high frequency heart rate variability between baseline and 180 days after enrollment.
Change in inflammatory marker high-sensitivity C-reactive protein | 180 days after enrollment
  Change in high sensitivity C-reactive protein (hsCRP) between baseline and 180 days after enrollment.
Change in inflammatory marker interleukin-6 | 180 days after enrollment
  Change in interleukin-6 (IL6) between baseline and 180 days post-enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Meadows, M.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
After the study period, all identifiers will be removed from data and specimen, but the de-identified dataset free of PHI specifiers will be uploaded to a data sharing service.
Time Frame: Beginning 1 year after publication with no end date
Access Criteria: Data will be available in a data sharing repository